CLINICAL TRIAL: NCT02312284
Title: Observational Study on the Patients With Rectal Cancer: Experience From Cancer Hospital, Chinese Academy of Medical Sciences 2000-2010
Brief Title: Observational Study on the Patients With Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., MD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CAMS 14-122/912
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Rectal Cancer; Adjuvant Chemoradiotherapy; Neoadjuvant Chemoradiotherapy; Adjuvant Chemotherapy; Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Radiotherapy/Chemoradiotherapy: Pre- or postoperative or palliative radiotherapy/chemoradiotherapy based on 5-fluorouracil or Capecitabine +/-Oxaliplatin
- Surgery: Transabdominal resection or transanal excision
- Chemotherapy: Pre- or postoperative chemotherapy including 5-fluorouracil/leucovorin with oxaliplatin, Capecitabine, etc

SUMMARY:
The aim of this observational study is to retrospectively collect current survival data for 3995 primary rectal cancer patients who were extracted from 5097 rectal cancer patients admitted in Cancer Hospital, Chinese Academy of Medical Sciences from January 2000 to December 2010. Moreover, based on a Cox model, we want to develope a nomogram that predicts local recurrence, distant metastases, and survival for patients with rectal cancer treated with pre- or postoperative chemoradiotherapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Aged older than 18 years
* American Joint Committee on Cancer (six edition) stage I through IV disease
* Received either transabdominal resection, transanal excision, preoperative radiotherapy or chemoradiotherapy
* Had the histologic subtypes adenocarcinoma (not otherwise specified, mucinous or mucin-producing, mixed cell or with mixed subtypes, tubular, and papillary)

Exclusion Criteria:

* Had the histologic subtypes squamous cell carcinoma, carcinoid, neuroendocrine tumor, small cell carcinoma, leiomyosarcoma, sarcoma, gastrointestinal stromal sarcoma, melanoma, carcinosarcoma, rhabdoid tumors, or malignant peripheral nerve sheet tumors
* Only receive palliative surgery such as colostomy, sigmoidostomy
* Received palliative radiotherapy or chemoradiotherapy for metastatic disease
* With unresectable distant metastasis in liver, lung, bone, central nervous system , or peritoneal transplantation
* Had no detailed medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical, pathological and routine laboratory characteristics for 3995 patients were extracted from 5097 patients with rectal cancer treated in Cancer Hospital, Chinese Academy of Medical Sciences from 2000 to 2010.The clinical data were reviewed and a prediction nomogram based on the Cox proportional hazards model were developed.
Sampling Method: Non-Probability Sample
Enrollment: 3995 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5-10 years
Cancer-specific survival | 5-10 years
Locoregional recurrence free survival | 5-10 years
Distant metastasis free survival | 5-10 years

SECONDARY OUTCOMES:
Chemotherapy/Radiotherapy/Chemoradiotherapy toxicities | the duration of hospital stay (an expected average of 6 weeks for chemoradiotherapy and 4-6 months for chemotherapy), as well as within 30 days after completion of the treatment and all the follow-up time
  Chemotherapy toxicities are evaluated by NCI-CTC version 3.0 and radiotherapy toxicities are graded using the RTOG/EORTC Radiation Morbidity Scoring Schema.
Surgery complication | within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China

REFERENCES:
- [Derived] Liu W, Jin J, Li Y, Wang S, Song Y, Liu Y, Wang W, Ren H, Fang H, Li N, Tang Y, Wang X, Tang Y, Lu N, Xiao Q, Feng Y, Wang J, Deng L, Jing H, Liu X, Yu Z. [Radical surgery combined with adjuvant radiotherapy for elderly patients aged over 75 years with stage II( or III( rectal cancer: a retrospective study from a single center]. Zhonghua Wei Chang Wai Ke Za Zhi. 2018 Jun 25;21(6):654-659. Chinese. PMID 29968240